CLINICAL TRIAL: NCT04297358
Title: Hyperbaric Oxygen Treatment in Chronic Stroke a Feasibility Study
Brief Title: Hyperbaric Oxygen in Patients Who Had a Stroke
Acronym: HOST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hyperbaric Center Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02131
Record Dates: First submitted 2020-02-26; First posted 2020-03-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Hyperbaric Oxygen
Keywords: Hyperbaric Oxygen; Completed Stroke; Feasibility; Prospective
MeSH Terms: conditions — Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stroke patients (Experimental): 40 consecutive sessions of hyperbaric oxygen will be administered at a pressure of 2 absolute atmosphere (ATA) to 10 patients. If there are drop outs, recruitment will be continued until a total of 10 patients with at least 30 sessions.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — 40 consecutive (5/7) sessions of hyperbaric oxygen

SUMMARY:
Prospective clinical assessment of 40 Hyperbaric Oxygen (HBO) treatments in 10 completed stroke patients.

DETAILED DESCRIPTION:
10 patients having suffered a stroke and having being rehabilitated will be treated with 40 consecutive Hyperbaric Oxygen Treatment (HBOT) after a minimal delay of 3 months after stroke. They will be neurologically assessed before and 3 months after HBOT. Rivermead mobility index will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic cortical stroke in chronic stage (≥ 3 months) with residual motor deficits confirmed by imaging with brain CT scan and/or brain MRI

Informed consent

Exclusion Criteria:

* Neurological issue:

  * inability to understand the informed consent form
  * Hemiplegia
* Hyperbaric issue:

  * Claustrophobia
  * inability to put on face mask
  * uncontrolled epilepsy
  * dementia or psychological disturbance
  * previous pneumothorax
  * pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in National Institutes of Health Stroke Scale (NIHSS score) | Change from Baseline NIHSS Score at 3 months
  Neurological assessment before and after HBOT. Composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0 (0 is better).
Change in Rivermead mobility index (RMI) at 2 weeks | Change from Baseline RMI at 2 weeks
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.
Change in Rivermead mobility index (RMI) at 4 weeks | Change from Baseline RMI at 4 weeks
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.
Change in Rivermead mobility index (RMI) at 6 weeks | Change from Baseline RMI at 6 weeks
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.
Change in Rivermead mobility index (RMI) at 8 weeks | Change from Baseline RMI at 8 weeks
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.
Change in Rivermead mobility index (RMI) at 1 month | Change from Baseline RMI at 1 month
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.
Change in Rivermead mobility index (RMI) at 3 months | Change from Baseline RMI at 3 months
  Mobility scale used in neurological rehabilitation. All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15 (15 is better). Changes are evaluated every two weeks for a total of 8 weeks (every 10 sessions of HBOT), than after 1 and 3 months.

SECONDARY OUTCOMES:
Tympanic damage | From date of Start of HBOT until the date of End of HBOT
  Digital photography before and after each daily HBOT session, that means before and after each compression/decompression in the hyperbaric chamber, to detect any ear lesion.
Change in Visual Acuity | Change from Baseline Visual Acuity at 3 months
  Snellen chart. Visual acuity test from a distance of 6m. 1 is normal vision, 0 is blindness. Each eye is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gelsomino, med pract, Principal Investigator — Druckkammerzentrum Basel
Locations (1):
- Druckkammerzentrum Basel, Basel, Switzerland